CLINICAL TRIAL: NCT04670887
Title: A Prospective Multicenter Trial Comparing Surgery Versus Active Surveillance In Patients With Bosniak 3 Renal Cystic Masses, A NoRenCa And FinnKidney Study
Brief Title: Comparison of Surgery and Active Surveillance in the Treatment of Bosniak III Renal Cysts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Harry Nisén, Adjunct professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/1556/2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-12

CONDITIONS: Cystic Renal Disease; Kidney Cancer; Surgery
Keywords: Bosniak classification; Active surveillance; Renal cystic mass; Cystic renal cell carcinoma
MeSH Terms: conditions — Kidney Diseases, Cystic; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate surgery (Active Comparator): Patients undergo excision of a renal mass by partial or radical nephrectomy and will be followed by UISS risk classification.
  Interventions: Procedure: Immediate surgery
- Active surveillance (Active Comparator): Patients enter active surveillance protocol. Delayed surgery on active surveillance will be recommended if progression from Bosniak 3 to 4 or a solid mass is noted on imaging by radiologist
  Interventions: Procedure: Delayed surgery

INTERVENTIONS:
Procedure: Delayed surgery — Delayed surgery is performed if cystic mass radiologically upgrades into Bosniak 4 or solid mass in the active surveillance.
  Arms: Active surveillance
Procedure: Immediate surgery — Partial or radical nephrectomy is performed as treatment of Bosniak 3 cystic mass
  Arms: Immediate surgery

SUMMARY:
The incidence of renal cysts is rising due to increased abdominal imaging. Renal complicated cysts have been traditionally classified according to the Bosniak classification, which distinguishes cystic masses by specific features of walls and septa. The categories I and II are benign and class IIF most probably benign but needs a short radiological follow-up. Categories III and IV have been traditionally operated due to the increased risk of renal cell carcinoma. However, recently published studies show that approximately 50% of the operated Bosniak III cystic masses are benign, which means that half of the cases are overtreated by surgery. It has also been shown that surgical pathology of stable Bosniak IIF cysts is malignant in less than 1%, while the cysts, which are upgraded to higher Bosniak classes will show malignant surgical pathology in 85%. So far, there is lack of prospective data on active surveillance in Bosniak III cystic masses.

The aim of the study is to compare active surveillance and surgery in patients with Bosniak III renal cystic masses. Patients will be randomized in active surveillance or immediate surgical excision of a cystic mass. In the active surveillance group, patients are followed according to the study protocol for 10 years and treated with delayed surgery if the cystic mass upgrades into Bosniak IV/solid, becomes symptomatic or grows over a preclassified threshold. The primary objective is to compare surgical pathology between patients treated with immediate surgery versus delayed surgery.

According to recent retrospective data, active surveillance of Bosniak III cystic masses is reasonable and oncologically safe. Therefore a prospective randomized controlled trial is needed to get high level evidence to support a change in the treatment strategy. The study may significantly reduce unnecessary operations performed in patients with Bosniak III cystic masses.

ELIGIBILITY:
Inclusion Criteria:

* A sporadic single CM of Bosniak 3 according to the Bosniak Classification v.2019 is diagnosed with CT or MRI
* Maximal diameter of CM 10-70 mm
* Age ≥50 years
* ECOG performance status <2
* Life expectancy ≥5 years
* Patient is fit to undergo surgery and AS.
* Patient understands a national language or English
* Signed informed consent

Exclusion Criteria:

* Genetic syndromes associated with RCC
* Previously or simultaneously diagnosed and pathologically verified RCC
* Previously or simultaneously radiographically identified solid mass or CM of Bosniak 3/4 with diameter ≥10mm
* The target CM of Bosniak 3 has progressed in sequential imaging from Bosniak 1-2F
* Presence of radiographic findings which are suspect for nodal or distant metastatic disease
* Symptomatic CM
* Kidney insufficiency (GFR<55 ml/min/1,73m2)
* Patients who have contraindications for both CT and MRI imaging. . Anatomically solitary kidney

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2024-01-11 (Estimated); Study Completion 2036-01-11 (Estimated)

PRIMARY OUTCOMES:
Malignancy rate in surgical pathology | From date of randomization until the date of surgery, assessed up to 120 months

SECONDARY OUTCOMES:
Cancer specific survival | From date of randomization until the date of death due to renal cancer, assessed up to 120 months
Progression-free survival | From date of randomization until the date of first documented progression, assessed up to 120 months
Overall survival | From date of randomization until the date of death from any cause, assessed up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Harry Nisén, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: Requests are reviewed by the steering committee.